CLINICAL TRIAL: NCT02140684
Title: Exhaled Nitric Oxide in Asthma Management: a Retrospective Real-life Observational Evaluation of the Use of Exhaled Nitric Oxide Measurements for Asthma Management in a UK Primary Care Population
Brief Title: Exhaled Nitric Oxide in Asthma Management
Status: Suspended | Type: Observational
Why Stopped: suspended due to lack of data.
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Aerocrine AB (Industry)
Responsible Party: Principal Investigator, David Price, Prof., MD, David Price, Research in Real-Life Ltd
Other Study IDs: 009/12
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: Real-world; observational; Nitric oxide; Inhaled corticosteroid; UK
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- eNO monitoring: Patients undergoing eNO monitoring at the index prescription date
  Interventions: Device: eNO monitoring
- No eNO monitoring

INTERVENTIONS:
Device: eNO monitoring — Patient undergoing review with eNO monitored using either NIOX MINO® and NIOX Flex®
  Groups: eNO monitoring

SUMMARY:
This study will compare the absolute and relative effectiveness of managing real-life asthma with and without the use of NIOX MINO® and NIOX Flex® to measure exhaled nitric oxide (eNO) as a marker of underlying airway inflammation to guide appropriate management. As exhaled nitric oxide responds rapidly to environmental changes and can act as a marker of underlying inflammation it is proposed that incorporating eNO monitoring into routine asthma management treatment allows strategies to be more accurately tailored to the patients needs, increasing the probability of good asthma control.

ELIGIBILITY:
Inclusion Criteria:

1. Aged: 6-80 years
2. Evidence of active asthma (diagnostic code and/or ≥6 prescriptions for asthma therapy at any time in their records)
3. Evidence of current asthma treatment (≥2 asthma prescriptions during baseline year and outcome year)
4. Have at least one year of up-to-standard (UTS) baseline data and at least one year of UTS outcome data (following the IPD)

Exclusion Criteria:

1. Had a COPD read code at any time; and/or
2. Had any chronic respiratory disease, except asthma, at any time; and/or
3. Patients on maintenance oral steroids during baseline year
4. Smoker or ex-smoker aged over 60

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asthma patients who either:
  * Use eNO monitoring in their asthma management
  * Do not use eNO monitoring
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Severe Exacerbation Rate | One Year Outcome Period
  Where exacerbations are defined as an occurrence of:
  Unscheduled hospital admissions / Emergency Room attendance for asthma, OR Use of acute courses of oral steroids
Proxy Asthma Control | One year outcome period
  1. No recorded hospital attendance for asthma, including admission, Emergency Room (ER) attendance or Out-Patient Department (OPD) attendance, AND
  2. No prescriptions for acute courses of oral steroids, AND
  3. No GP consultations, hospital admissions or ER attendance for lower respiratory tract infections (LRTI) requiring antibiotics.

SECONDARY OUTCOMES:
Asthma Control (including SABA) | One year outcome
  Proxy asthma control (defined above), including the absence of average daily prescribed dose of ≤200mcg salubtamol / ≤500mcg terbutaline
Respiratory-related hospitalisations and referrals | One year outcome period
  Mean number of respiratory-related hospitalisations and referrals per patient during the outcome year

CONTACTS AND LOCATIONS:
Locations (1):
- Research in Real Life, Cambridge, United Kingdom

REFERENCES:
- [Background] Clancy RM, Amin AR, Abramson SB. The role of nitric oxide in inflammation and immunity. Arthritis Rheum. 1998 Jul;41(7):1141-51. doi: 10.1002/1529-0131(199807)41:73.0.CO;2-S. No abstract available. PMID 9663469
- [Background] Baraldi E, Carra S, Dario C, Azzolin N, Ongaro R, Marcer G, Zacchello F. Effect of natural grass pollen exposure on exhaled nitric oxide in asthmatic children. Am J Respir Crit Care Med. 1999 Jan;159(1):262-6. doi: 10.1164/ajrccm.159.1.9804063. PMID 9872848
- [Background] Piacentini GL, Bodini A, Costella S, Vicentini L, Peroni D, Zanolla L, Boner AL. Allergen avoidance is associated with a fall in exhaled nitric oxide in asthmatic children. J Allergy Clin Immunol. 1999 Dec;104(6):1323-4. doi: 10.1016/s0091-6749(99)70031-x. No abstract available. PMID 10589019
- [Background] Bukstein D, Luskin AT, Brooks EA. Exhaled nitric oxide as a tool in managing and monitoring difficult-to-treat asthma. Allergy Asthma Proc. 2011 May-Jun;32(3):185-92. doi: 10.2500/aap.2011.32.3449. Epub 2011 Apr 8. PMID 21477457
- See also: RIRL company webpage — http://www.rirl.org/